CLINICAL TRIAL: NCT06325488
Title: Fibrosis, Inflammation, Oxygenation of Renal Tissue In FabrY Disease
Acronym: FORTIFY
Status: Recruiting | Type: Observational
Sponsor: Caroline Michaela Kistorp (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Caroline Michaela Kistorp, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-23035668
Record Dates: First submitted 2024-02-14; First posted 2024-03-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Fabry Disease; Chronic Kidney Diseases
Keywords: Oxygenation; Inflammation; Fibrosis
MeSH Terms: conditions — Fabry Disease; Renal Insufficiency, Chronic; Inflammation; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Fabry Disease and impaired kidney function: Participants included in this group
  * 18 years of age or above
  * Fabry Disease as verified by genetic analysis prior to inclusion
  * Impaired kidney function according to the KDIGO classification (UACR ≥ 30 mg/g and eGFR < 60 ml/min/1.73m2 [≥ CKD G3a/A2])
- Patients with Fabry Disease and normal kidney function: Participants included in this group
  * 18 years of age or above
  * Fabry Disease as verified by genetic analysis prior to inclusion
  * Normal kidney function according to the KDIGO classification (UACR < 30 mg/g and eGFR ≥ 60 will be included [≤ CKD G2/A1])
- Healthy controls: Participants included in this group
  * 18 years of age or above
  * Normal kidney function according to the KDIGO classification (UACR < 30 mg/g and eGFR ≥ 60 will be included [≤ CKD G2/A1])
  Furthermore, healthy controls are excluded
  * Suspected of Fabry Disease or verified by genetic analysis
  * Related to a patient with Fabry Disease
  * Have cancer with an expected influence on life expectancy
  * Known apoplexia cerebri, heart failure or established kidney disease
  * Recently initiated or have had recent changes in antihypertensive medication (within 3 months)

SUMMARY:
The overall objective of this study is to investigate Fabry-associated renal organ involvement by using a novel magnetic resonance imaging (MRI) approach, focusing on changes in renal oxygen levels by blood oxygenation-level dependent (BOLD) imaging. Furthermore, to correlate renal oxygenation to the phenotypic presentation of patients with Fabry-associated nephropathy regarding circulating and imaging-derived biomarkers of kidney inflammation, fibrosis and injury as compared with healthy age- and sex-matched controls.

The study will achieve this by:

1) Using a non-invasive, contrast-free MRI protocol focusing on parameters of oxygenation, inflammation, fibrosis, and injury in the kidney.

2) Using an extensive, in-depth biomarker blood panel to investigate the pathological pathways associated with Fabry disease and Fabry-associated nephropathy.

DETAILED DESCRIPTION:
From attached protocol:

Introduction Fabry disease is a rare X-linked lysosomal disorder caused by mutations in the gene encoding the enzyme alpha-galA, an essential enzyme for normal cellular function. The enzyme deficiency causes progressive accumulation of glycosphingolipids, especially globotriaosylceramide (Gb3) in virtually all organs, leading to dysfunction and eventually leading to organ failure. Although, Fabry disease is caused by an X-linked genetic mutation and the clinical implication among men with a classic phenotype are most severe, Fabry disease affects both males and females. Men with a non-classic phenotype and females present with a more heterogenous degree of organ involvement, however, these patients remain at increased risk of multisystem organ involvement and must be attend extensive screening, evaluated repeatedly in order to decide when and who are in need of treatment. However, as evident in patients with the several known genotypes, which presents with no or very low alpha-galA-activity and develop early multi-organ involvement, one of the complication of greatest prognostic impact is an early involvement of the kidney.

Fabry nephropathy Although, the etiology of kidney affection in Fabry disease in general is well established, the actual mechanisms of progression - and thus the targets of therapeutic approach - are largely unknown. Fabry nephropathy is characterized by the accumulation of Gb3 deposition in podocytes, epithelial cells and endothelial cells throughout the tubules, where kidney biopsies suggest healthy, functioning tissue is substituted with reparative diffuse fibrosis. Indeed, evidence shows a direct association between Gb3 accumulation and both a decline in renal glomerular filtration rate and an increase in urinary albumin excretion - both clinically validated biomarkers of kidney injury and decline in function. Given Gb3 accumulation in Fabry disease accounts for less than 5% of the total tissue volume at maximum, the disproportionate and devastating effects observed have led to the proposal of Gb3 having additional effects beyond mere storage. Oxidative stress, endothelial dysfunction, and inflammation have been proposed as important mechanisms induced directly or indirectly by Gb3 accumulation, resulting in increased cell-death of functioning glomeruli with unamenable, reparative fibrosis as a result. Furthermore, certain cells seems more susceptible to injury and less susceptible to the benefits expected from Fabry-specific treatment; an important example being renal podocytes.

Fabry nephropathy and Magnetic Resonance Imaging Renal hypoxia is now considered to play a key role in the development of chronic kidney disease (CKD). Using a novel contrast-free, non-invasive magnetic resonance imaging (MRI), our collaborative partners have reported renal hypoxia in subjects with type I diabetes and pathological urinary albumin/creatinine ratio (UACR) levels. Recent advances in MRI thus, enables us to investigate the pathological mechanisms underlining Fabry nephropathy by non-invasively measurements of oxygenation, inflammation and fibrosis. The kidney's oxidative capacity evaluated by R2*-related blood oxygenation level-dependent (BOLD) MRI has been validated as a parameter of renal cortical and medullar oxygen-partial pressure. Furthermore, changes in dynamic R2*-signaling have been validated as a non-invasive, contrast-free measure of renal oxygenation capacity, which becomes reduced with presence of chronic kidney disease. Concurrently, arterial spin labelling (ASL) is able to provide a reliable measure of total blood flow as well as regional blood flow in the renal artery and the kidney. Finally, the inflammatory and fibrotic burden can be elucidated upon by diffusion-weighted sequences and native T1-mapping. Therefore, this novel method provides information on kidney-specific shift in energetic oxygen-dependent capacity, ongoing inflammation, and accumulation of fibrosis, with changes not only portraying key aspects of kidney physiology, but changes expected to elucidate on the pathophysiology forming the very basis of Fabry nephropathy.

While the recent advances in imaging present a unique possibility for early detection of Fabry nephropathy, there is a need for validation against clinically established biomarkers of risk such as pathologically increased UACR - currently the greatest predictor of progressive loss of glomerular function in regards to end-stage renal disease in general and in Fabry nephropathy. Pathological UACR levels is considered the first clinical sign of Fabry nephropathy, with an estimated prevalence of 50% among men aged 35 years. Even among women, which often less severely afflicted, up to 40% develop proteinuria and 15% experience a clinically significant renal event, thus, the prognostic importance of increased UACR in Fabry disease is evident. Therefore, UACR levels is the key clinical parameter of Fabry nephropathy as recommended in guidelines.

ELIGIBILITY:
Fabry patients:

Inclusion Criteria:

* Male and female individuals (≥18 years of age)
* Able to give informed consent

Exclusion Criteria:

* Any contraindication for magnetic resonance imaging according to standard checklist used in clinical routine, including claustrophobia or metallic foreign bodies, metallic implants, internal electrical devices, or permanent makeup/tattoos that cannot be declared MR compatible.
* Pregnancy

Control group Inclusion criteria

* Male and female individuals (≥18 years of age)
* Able to give informed consent Exclusion criteria
* A genetically-verified diagnosis of Fabry disease.
* Family member to a patient with a genetically-verified diagnosis of Fabry disease
* Cancer expected to influence life expectancy.
* Known heart failure, previous apoplexia or previously established kidney disease.
* Initiation or change of antihypertensive therapy within 3 months of enrolment
* Renal impairment as depicted by the CKD-EPI classification (≥ CKD G2/A1)
* Any contraindication for MRI according to standard checklist used in clinical routine, including claustrophobia or metallic foreign bodies, metallic implants, internal electrical devices, or permanent makeup/tattoos that cannot be declared MR compatible.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with Fabry disease (n=40) - previously established by genetic testing - are to be grouped according to the presence of renal impairment as defined by the KDIGO criteria.
  A group of controls with no renal impairment are to act as healthy controls.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Renal hypoxia (Fabry patients according to renal impairment) | At baseline
  A between-group difference in renal hypoxia (R*) evaluated by BOLD MRI when comparing the groups of patients with Fabry disease.

SECONDARY OUTCOMES:
Renal hypoxia (Fabry patient vs controls) | At baseline
  A between-group difference in renal hypoxia (R*) evaluated by BOLD MRI when comparing patients with Fabry disease irrespective of renal impairment with the control group.
Renal cortical perfusion (Fabry vs. controls) | At baseline
  A between-group difference in perfusion of the renal medulla (mL/100g/min) when comparing groups with Fabry disease patients with the control group
Renal medullar perfusion (Fabry vs. controls) | At baseline
  A between-group difference in renal blood flow (mL/min) when comparing groups with Fabry disease patients with the control group.
Renal inflammation (Fabry vs. controls) | At baseline
  A between-group difference in native T1 (ms) when comparing groups with Fabry disease patients with the control group.
Renal fibrosis (Fabry vs. controls) | At baseline
  A between-group difference in diffusion-weigthed signaling when comparing groups with Fabry disease patients with the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Kistorp, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to national legistlative restrictions, unrestricted access to individual participant data is not possible. However, data exchange will be possible upon reasonable request under the assurance of data-management in accordance with Danish law.

REFERENCES:
- [Background] Waldek S, Patel MR, Banikazemi M, Lemay R, Lee P. Life expectancy and cause of death in males and females with Fabry disease: findings from the Fabry Registry. Genet Med. 2009 Nov;11(11):790-6. doi: 10.1097/GIM.0b013e3181bb05bb. PMID 19745746
- [Background] Wanner C, Germain DP, Hilz MJ, Spada M, Falissard B, Elliott PM. Therapeutic goals in Fabry disease: Recommendations of a European expert panel, based on current clinical evidence with enzyme replacement therapy. Mol Genet Metab. 2019 Mar;126(3):210-211. doi: 10.1016/j.ymgme.2018.04.004. Epub 2018 Apr 11. No abstract available. PMID 29724657
- [Background] Najafian B, Tondel C, Svarstad E, Gubler MC, Oliveira JP, Mauer M. Accumulation of Globotriaosylceramide in Podocytes in Fabry Nephropathy Is Associated with Progressive Podocyte Loss. J Am Soc Nephrol. 2020 Apr;31(4):865-875. doi: 10.1681/ASN.2019050497. Epub 2020 Mar 3. PMID 32127409
- [Background] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, Feliciani C, Shankar SP, Ezgu F, Amartino H, Bratkovic D, Feldt-Rasmussen U, Nedd K, Sharaf El Din U, Lourenco CM, Banikazemi M, Charrow J, Dasouki M, Finegold D, Giraldo P, Goker-Alpan O, Longo N, Scott CR, Torra R, Tuffaha A, Jovanovic A, Waldek S, Packman S, Ludington E, Viereck C, Kirk J, Yu J, Benjamin ER, Johnson F, Lockhart DJ, Skuban N, Castelli J, Barth J, Barlow C, Schiffmann R. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016 Aug 11;375(6):545-55. doi: 10.1056/NEJMoa1510198. PMID 27509102
- [Background] Jehn U, Bayraktar S, Pollmann S, Van Marck V, Weide T, Pavenstadt H, Brand E, Lenders M. alpha-Galactosidase a Deficiency in Fabry Disease Leads to Extensive Dysregulated Cellular Signaling Pathways in Human Podocytes. Int J Mol Sci. 2021 Oct 20;22(21):11339. doi: 10.3390/ijms222111339. PMID 34768768
- [Background] Linhart A, Elliott PM. The heart in Anderson-Fabry disease and other lysosomal storage disorders. Heart. 2007 Apr;93(4):528-35. doi: 10.1136/hrt.2005.063818. No abstract available. PMID 17401074
- [Background] Yogasundaram H, Kim D, Oudit O, Thompson RB, Weidemann F, Oudit GY. Clinical Features, Diagnosis, and Management of Patients With Anderson-Fabry Cardiomyopathy. Can J Cardiol. 2017 Jul;33(7):883-897. doi: 10.1016/j.cjca.2017.04.015. Epub 2017 May 4. PMID 28668140
- [Background] Eikrem O, Skrunes R, Tondel C, Leh S, Houge G, Svarstad E, Marti HP. Pathomechanisms of renal Fabry disease. Cell Tissue Res. 2017 Jul;369(1):53-62. doi: 10.1007/s00441-017-2609-9. Epub 2017 Apr 12. No abstract available. PMID 28401309
- [Background] Ravarotto V, Simioni F, Carraro G, Bertoldi G, Pagnin E, Calo LA. Oxidative Stress and Cardiovascular-Renal Damage in Fabry Disease: Is There Room for a Pathophysiological Involvement? J Clin Med. 2018 Nov 2;7(11):409. doi: 10.3390/jcm7110409. PMID 30400144
- [Background] Sanchez-Nino MD, Carpio D, Sanz AB, Ruiz-Ortega M, Mezzano S, Ortiz A. Lyso-Gb3 activates Notch1 in human podocytes. Hum Mol Genet. 2015 Oct 15;24(20):5720-32. doi: 10.1093/hmg/ddv291. Epub 2015 Jul 23. PMID 26206887
- [Background] Ravarotto V, Carraro G, Pagnin E, Bertoldi G, Simioni F, Maiolino G, Martinato M, Landini L, Davis PA, Calo LA. Oxidative stress and the altered reaction to it in Fabry disease: A possible target for cardiovascular-renal remodeling? PLoS One. 2018 Sep 27;13(9):e0204618. doi: 10.1371/journal.pone.0204618. eCollection 2018. PMID 30261035
- [Background] Fall B, Scott CR, Mauer M, Shankland S, Pippin J, Jefferson JA, Wallace E, Warnock D, Najafian B. Urinary Podocyte Loss Is Increased in Patients with Fabry Disease and Correlates with Clinical Severity of Fabry Nephropathy. PLoS One. 2016 Dec 16;11(12):e0168346. doi: 10.1371/journal.pone.0168346. eCollection 2016. PMID 27992580
- [Background] Selby NM, Blankestijn PJ, Boor P, Combe C, Eckardt KU, Eikefjord E, Garcia-Fernandez N, Golay X, Gordon I, Grenier N, Hockings PD, Jensen JD, Joles JA, Kalra PA, Kramer BK, Mark PB, Mendichovszky IA, Nikolic O, Odudu A, Ong ACM, Ortiz A, Pruijm M, Remuzzi G, Rorvik J, de Seigneux S, Simms RJ, Slatinska J, Summers P, Taal MW, Thoeny HC, Vallee JP, Wolf M, Caroli A, Sourbron S. Magnetic resonance imaging biomarkers for chronic kidney disease: a position paper from the European Cooperation in Science and Technology Action PARENCHIMA. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii4-ii14. doi: 10.1093/ndt/gfy152. PMID 30137584
- [Background] Pruijm M, Milani B, Burnier M. Blood Oxygenation Level-Dependent MRI to Assess Renal Oxygenation in Renal Diseases: Progresses and Challenges. Front Physiol. 2017 Jan 5;7:667. doi: 10.3389/fphys.2016.00667. eCollection 2016. PMID 28105019
- [Background] Heyman SN, Khamaisi M, Rosen S, Rosenberger C. Renal parenchymal hypoxia, hypoxia response and the progression of chronic kidney disease. Am J Nephrol. 2008;28(6):998-1006. doi: 10.1159/000146075. Epub 2008 Jul 18. PMID 18635927
- [Background] Inoue T, Kozawa E, Okada H, Inukai K, Watanabe S, Kikuta T, Watanabe Y, Takenaka T, Katayama S, Tanaka J, Suzuki H. Noninvasive evaluation of kidney hypoxia and fibrosis using magnetic resonance imaging. J Am Soc Nephrol. 2011 Aug;22(8):1429-34. doi: 10.1681/ASN.2010111143. Epub 2011 Jul 14. PMID 21757771
- [Background] Pruijm M, Mendichovszky IA, Liss P, Van der Niepen P, Textor SC, Lerman LO, Krediet CTP, Caroli A, Burnier M, Prasad PV. Renal blood oxygenation level-dependent magnetic resonance imaging to measure renal tissue oxygenation: a statement paper and systematic review. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii22-ii28. doi: 10.1093/ndt/gfy243. PMID 30137579
- [Background] Laursen JC, Sondergaard-Heinrich N, Haddock B, Rasmussen IKB, Hansen CS, Larsson HBW, Groop PH, Bjornstad P, Frimodt-Moller M, Andersen UB, Rossing P. Kidney oxygenation, perfusion and blood flow in people with and without type 1 diabetes. Clin Kidney J. 2022 May 20;15(11):2072-2080. doi: 10.1093/ckj/sfac145. eCollection 2022 Nov. PMID 36825032
- [Background] Wilcox WR, Oliveira JP, Hopkin RJ, Ortiz A, Banikazemi M, Feldt-Rasmussen U, Sims K, Waldek S, Pastores GM, Lee P, Eng CM, Marodi L, Stanford KE, Breunig F, Wanner C, Warnock DG, Lemay RM, Germain DP; Fabry Registry. Females with Fabry disease frequently have major organ involvement: lessons from the Fabry Registry. Mol Genet Metab. 2008 Feb;93(2):112-28. doi: 10.1016/j.ymgme.2007.09.013. Epub 2007 Nov 26. PMID 18037317
- [Background] Deegan PB, Baehner AF, Barba Romero MA, Hughes DA, Kampmann C, Beck M; European FOS Investigators. Natural history of Fabry disease in females in the Fabry Outcome Survey. J Med Genet. 2006 Apr;43(4):347-52. doi: 10.1136/jmg.2005.036327. Epub 2005 Oct 14. PMID 16227523
- [Background] Warnock DG, Thomas CP, Vujkovac B, Campbell RC, Charrow J, Laney DA, Jackson LL, Wilcox WR, Wanner C. Antiproteinuric therapy and Fabry nephropathy: factors associated with preserved kidney function during agalsidase-beta therapy. J Med Genet. 2015 Dec;52(12):860-6. doi: 10.1136/jmedgenet-2015-103471. Epub 2015 Oct 21. PMID 26490103
- [Background] Hughes DA, Aguiar P, Deegan PB, Ezgu F, Frustaci A, Lidove O, Linhart A, Lubanda JC, Moon JC, Nicholls K, Niu DM, Nowak A, Ramaswami U, Reisin R, Rozenfeld P, Schiffmann R, Svarstad E, Thomas M, Torra R, Vujkovac B, Warnock DG, West ML, Johnson J, Rolfe MJ, Feriozzi S. Early indicators of disease progression in Fabry disease that may indicate the need for disease-specific treatment initiation: findings from the opinion-based PREDICT-FD modified Delphi consensus initiative. BMJ Open. 2020 Oct 10;10(10):e035182. doi: 10.1136/bmjopen-2019-035182. PMID 33039984

DOCUMENTS (2):
  • Study Protocol (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT06325488/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT06325488/SAP_001.pdf